CLINICAL TRIAL: NCT02970617
Title: Are Last Impressions Lasting Impressions? Intervention of Ringing a Bell at the End of Cancer Treatment
Brief Title: Ringing a Bell on the Final Day of Radiation Therapy in Improving the Memory of Distress in Cancer Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern California (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: OS-15-15; NCI-2016-01259 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); OS-15-15 (Other: USC / Norris Comprehensive Cancer Center); P30CA014089 (NIH)
Record Dates: First submitted 2016-11-15; First posted 2016-11-22 (Estimated); Last update posted 2025-10-07 (Actual); Status verified 2020-04

CONDITIONS: Distress; Malignant Neoplasm
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (no bell after final radiation) (Active Comparator): Patients undergo standard of care radiation therapy with or without chemotherapy.
  Interventions: Other: Questionnaire Administration
- Group B (ring bell after final radiation treatment) (Experimental): On the final day of standard of care radiation therapy, patients ring a bell in the clinic.
  Interventions: Other: Memory Intervention; Other: Questionnaire Administration

INTERVENTIONS:
Other: Memory Intervention — Ring bell after final radiation treatment
  Arms: Group B (ring bell after final radiation treatment)
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This clinical trial studies how well ringing a bell on the final day of radiation therapy works in improving the memory of distress in cancer patients. Ringing a bell on the final day of radiation therapy may improve the memory of how painful the treatment was.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine if the simple act of ringing a bell at the end of radiotherapy can improve the retrospective evaluation of distress due to radiotherapy and other prior cancer therapy.

SECONDARY OBJECTIVES:

I. To measure the severity of patients' memory of distress from cancer treatment.

II. To assess the relationship between anxiety to actual distress and to remembered distress.

III. To assess the relationship between optimism-pessimism personality to actual distress and to remembered distress.

IV. To assess patient's cognitive dissonance reduction to actual distress and to remembered distress.

OUTLINE: Patients are assigned to 1 of 2 groups.

GROUP A (No bell ringing): Patients undergo standard of care radiation therapy with or without chemotherapy.

GROUP B (Bell ringing): On the final day of standard of care radiation therapy, patients ring a bell in the clinic.

After completion of study, patients are followed up for 7 months.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of cancer
* Definitive radiation treatment with or without concurrent chemotherapy with curative intent; treatment prior to radiation therapy is acceptable (e.g. surgery, chemotherapy)
* Ability to understand and the willingness to sign a written informed consent; consents will be provided in English or Spanish
* Able to speak English or Spanish (questionnaires will be in English and Spanish)

Exclusion Criteria:

* Patients with either a malignant central nervous system (CNS)-primary cancer or with brain metastases; patients do not need to undergo brain imaging unless indicated per standard workup and management (e.g. advanced stage lung cancer receiving definitive therapy)
* Patients who will be receiving surgery or adjuvant chemotherapy within 1 month following radiation treatment
* Patients with widespread metastatic disease (> 3 distant metastases); patients with oligometastatic disease (=< 3 distant metastases) are allowed only if they are receiving definitive (curative) radiation therapy (RT) with or without chemotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2016-08-15 (Actual); Primary Completion 2018-11-15 (Actual); Study Completion 2018-11-15 (Actual)

PRIMARY OUTCOMES:
Distress memory scales as assessed by the 11-point Numeric Rating Scale | Up to 7 months
  Patient baseline characteristics and treatment will be summarized in groups A and B. Repeated measures analysis of variance (ANOVA) will be used to compare distress memory scales between patients in group A and group B. A mixed regression model will be used to examine the effect of ringing the bell on the last day of radiotherapy on distress memory scales when considering covariates such as baseline patient characteristics, cancer type, radiotherapy total dose and duration, baseline distress scale, analgesic medication, disease recurrence status, optimism/pessimism personality and anxiety.

SECONDARY OUTCOMES:
Anxiety level as assessed by Generalized Anxiety Disorder 7 scale | Up to 7 months
  Repeated measures ANOVA will be used to compare anxiety levels between patients in group A and group B. All p values will be two-sided at a significance level of 0.05.
Optimism-pessimism scores as assessed by the Life Orientation Test-Revised | Up to 7 months
  Repeated measures ANOVA will be used to compare optimisim-pessimism scores between patients in group A and group B. All p values will be two-sided at a significance level of 0.05.

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Williams, Principal Investigator — University of Southern California
Locations (1):
- USC / Norris Comprehensive Cancer Center, Los Angeles, California, United States